CLINICAL TRIAL: NCT03919838
Title: Effect of Probiotic Lactobacillus Salivarius and Cranberry on Oral Health of Children
Brief Title: Effect of Probiotic on Oral Health of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: NutroPharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KB/232/2016
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-06

CONDITIONS: Oral Disease
Keywords: probiotic; oral health; children
MeSH Terms: conditions — Mouth Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Participants will receive two lozenges containing probiotic bacteria and cranberry.
  Interventions: Dietary Supplement: Probiotics
- Placebo - No probiotics (Placebo Comparator): Participants will receive a control two lozenges containing no probiotic bacteria.
  Interventions: Dietary Supplement: Placebo - No probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — A half of the participants will be randomly allocated to the probiotics group. They will receive two probiotics lozenge before falling asleep for 8 weeks. Clinical examination will be conducted before study and after 8 weeks.
  Arms: Probiotics
Dietary Supplement: Placebo - No probiotics — A half of the participants will be randomly allocated to the placebo group. They will receive two no probiotics lozenge before falling asleep for 8 weeks. Clinical examination will be conducted before study and after 8 weeks.
  Arms: Placebo - No probiotics

SUMMARY:
The aim of the randomized, double-blind clinical trial with placebo is to answer the clinical question , or in children with diagnosed childhood early caries the use of L.salivarius and cranberry contained in NutroPharma lozenges will reduce new carious lesions and reduce the titre of the carcinogenic bacteria Streptococcus mutans, compared to the control group in which the placebo will be administered? The main end point will be to reduce the titre of cariogenic bacteria.

DETAILED DESCRIPTION:
Probiotic bacteria are used in the prevention and treatment of gastrointestinal diseases and infections, including the treatment of oral diseases. Probiotic bacteria can be found in saliva, plaque and adhering directly to the mucous membrane. They compete with cariogenic bacteria and pathogens of periodontal disease. Increased interest in probiotics means that attempts are being made to find new solutions regarding the methods of their administration. The use of probiotic bacteria brings beneficial health effects. Lactobacillus salivarius is a strain isolated from human milk. It is inactive (heat treatment) and therefore does not produce metabolites that can promote the formation of carious lesions in the mouth by lowering the mouth potential of hydrogen.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy children aged 3-6;
* recognized caries of early childhood, dmf> 1,
* lack of active caries and inflammation of the mouth
* colony forming unit CFU > 105 / ml Streptococcus mutans
* a minimum of one-month period from: the last antibiotic therapy, probiotic use, professional fluoride prophylaxis or supervised tooth brushing with fluoride preparations, the use of fluoride toothpaste, not using xylitol, written consent of parents / legal guardians for participation in research.

Exclusion Criteria:

* chronic diseases and chronically taken medicines in the past,
* planned change of residence during the year,
* age below 3 and above 6 years,
* healthy teeth, dmf = 0,
* colony forming unit CFU <105 / ml Streptococcus mutans
* Patient during antibiotic therapy, probiotic use, professional fluoride prophylaxis or supervised tooth brushing with fluoride preparations
* no toothpaste with fluoride
* using xylitol
* lack of written consent of parents / legal guardians for participation in research.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changing the titre of the carcinogenic bacteria Streptococcus mutans | 8 weeks
  During control tests saliva will be applied to the medium for identification and detailed quantification of S. mutans bacteria. After the incubation, the number of bacteria will be expressed - taking into account the degree of saliva dilution - as the number of colony-forming unit (CFU) in 1 ml of saliva.

CONTACTS AND LOCATIONS:
Locations (1):
- Dorota Olczak-Kowalczyk, Warsaw, Warsaw, 18 Miodowa Saint, Poland